CLINICAL TRIAL: NCT02476864
Title: Single-center, Open-label, Randomized, Two-treatment, Single-dose, Crossover Study in Healthy Subjects to Investigate the Biocomparison of the Adult and Pediatric Formulation of Macitentan
Brief Title: Comparison of the Pharmacokinetic Properties of Two Tablet Formulations of Macitentan in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AC-055-121; 2015-001623-23 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-06-22 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Subjects
Keywords: macitentan; biocomparison; safety
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Subjects receive treatment A in Period 1 followed by treatment B in Period 2 with a washout phase of 10 to 14 days between the two treatment periods
  Interventions: Drug: Treatment A (adult formulation); Drug: Treatment B (pediatric formulation)
- Sequence BA (Experimental): Subjects receive treatment B in Period 1 followed by treatment A in Period 2 with a washout phase of 10 to 14 days between the two treatment periods
  Interventions: Drug: Treatment A (adult formulation); Drug: Treatment B (pediatric formulation)

INTERVENTIONS:
Drug: Treatment A (adult formulation) — Single oral administration of one film-coated tablet containing 10 mg of macitentan as active substance and lactose, magnesium stearate, microcrystalline cellulose, povidone, sodium starch glycolate type A, polysorbate as inactive ingredients.The film coat contains titanium dioxide, talc, xanthan gum, polyvinyl alcohol, and soy lecithin.
  Other Names: Opsumit
Drug: Treatment B (pediatric formulation) — Single oral administration of two dispersible tablets, each containing 5 mg of macitentan as active ingredient and Mannitol delta polymorphic crystals, mannitol, isomalt, isomalt agglomerated, croscarmellose sodium, and magnesium stearate as inactive ingredients.

SUMMARY:
A study conducted in healthy adults to investigate if a new macitentan tablet leads to the same fate of macitentan in the body (time of onset, time of presence, amount in the blood) as the marketed macitentan tablet.

DETAILED DESCRIPTION:
The purpose of this study is to establish biocomparison of 2 types of tablets containing macitentan: a pediatric dispersible tablet and the adult film-coated tablet. A single oral dose of each tablet will be given to healthy subjects on 2 different periods separated by a washout phase of 10 to 14 days.

Biocomparison will be based on the comparison of the pharmacokinetic parameters of macitentan with the two types of tablets using specific statistical methods. The pharmacokinetic parameters will be considered equivalent if specific criteria defined in the study protocol are met.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy on the basis of the physical examination, vital signs (systolic and diastolic blood pressure, heart rate), 12-lead ECG, and laboratory tests performed at screening

Exclusion Criteria:

* History or clinical evidence of any disease and/or condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug
* Previous history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* History or clinical evidence of alcoholism or drug abuse within the 3 -year period prior to screening
* Excessive caffeine consumption
* Smoking within 3 months prior to screening and inability to refrain from smoking during the course of the study
* Previous treatment with any prescribed medications (including vaccines) or over-the counter medications within 2 weeks prior to first study drug administration
* Loss of 250 mL or more of blood within 3 months prior to screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic profile | From pre-dose to 216 hours post-dose
  Pharmacokinetic profile will be determined by the following parameters: Cmax (Maximum plasma concentration), tmax (Time to reach Cmax), t1/2 (Terminal half-life), AUC(0-t) (Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification), AUC(0-inf) (Area under the plasma concentration-time curve from zero to infinity)

OTHER OUTCOMES:
Incidence of adverse events | from baseline to Day 10-13 post-dose
  Number of adverse events and serious adverse events, including abnormal laboratory findings
ECG abnormalities | from baseline to to Day 10-13 post-dose
  ECG evaluation will be based on the cardiac rhythms measured using a standard 12-lead ECG device

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Sidharta, PharmD, PhD — Actelion